CLINICAL TRIAL: NCT00003100
Title: Metabolic Fate and Plasma Kinetics of Dietary Soy Isoflavones
Brief Title: Dietary Soy Isoflavones for the Prevention of Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000065832; UCMC-CHMC-91-5-3; NCI-P97-0117
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Soybean Proteins

INTERVENTIONS:
Dietary Supplement: soy isoflavones

SUMMARY:
RATIONALE: Eating a diet rich in soy foods appears to reduce the risk of some types of cancer. Isoflavones are compounds found in soy food that may prevent the development of cancer.

PURPOSE: Clinical trial to determine the most effective amount and type of soy isoflavones needed in the diets of healthy men and women to prevent cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of varying the dietary intake of soy nuts on plasma levels and urinary excretion of isoflavones. II. Determine the effects of different food composition, along with age and gender of subjects, on plasma levels and urinary excretion of isoflavones.

OUTLINE: This is a two part study. In part I; participants are stratified according to menopausal status. In part II; participants are stratified according to gender and age (under 50 vs. over 50). Part I - Study participants are given 3 different amounts of toasted soy nuts separated by one month intervals. The sequence in which each amount is given is randomized. Blood and urine samples are taken to measure isoflavone levels. Part II - Study participants are given toasted soy nuts, soy milk, and tempeh on separate occasions separated by one month intervals. The sequence of each food is randomized. Blood and urine samples are taken to measure isoflavone levels.

PROJECTED ACCRUAL: 10 women, 5 premenopausal and 5 postmenopausal, will be accrued for part I of the study. 80 subjects, 40 women and 40 men, will be accrued for part II.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Healthy women and men

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No chronic liver disease Renal: No chronic renal disease Cardiovascular: No chronic cardiovascular disease Pulmonary: No chronic pulmonary disease Other: No known allergy to soy proteins No consumption of soy protein within past week

PRIOR CONCURRENT THERAPY: Biologic therapy: No antibiotics within past 3 months Chemotherapy: Not specified Endocrine therapy: No oral contraceptive or hormone replacement therapy Radiotherapy: Not specified Surgery: Not specified Other: No medication likely to affect gastrointestinal, liver, or kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 1996-10

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Setchell, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio, United States